CLINICAL TRIAL: NCT01695018
Title: A Multicentral Prospective Study on Prediction of Malignant Progression of Oral Epithelial Dysplasia With p16 Methylation
Brief Title: Early Diagnosis of Oral Cancer by Detecting p16 Methylation
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Hongwei Liu, MD, PhD, Peking University School and Hospital of Stomatology, Peking University
Other Study IDs: PKUSSOM20120711
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Moderate Epithelial Dysplasia; Mild Epithelial Dysplasia
Keywords: oral epithelial dysplasia; p16 methylation; diagnostic reagents; early diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral mucosal biopsy tissues were formalin fixed , paraffin embedded , sliced and hematoxylin-eosin (HE) staining.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- p16 methylation positive: 48 patients with mild or moderate oral epithelial dysplasia containing methylated p16.
- p16 methylation negative: 104 patients with p16 mild or moderate oral epithelial dysplasia NOT containing methylated p16.

SUMMARY:
The purpose of this study is to verify the function of p16 methylation diagnostic reagents in early diagnosis of oral cancer.

DETAILED DESCRIPTION:
Background:Oral epithelial dysplasia (OED) is one of the common precancerous lesions among Chinese adults. To investigate the clinical predictive value of p16 methylation diagnostic reagents in the early diagnosis of oral cancer, the investigators carried out the prospective multi-center double-blind cohort study.

Methods:180 patients with histologically confirmed mild or moderate OED were included in the present study. The investigators using p16 methylation diagnostic reagents to analysis of the p16 methylation status in these patients. Building two follow-up queue by p16-methylated and p16-unmethylated. The Statistical analysis used SAS6.12 software. All P-values were two-sided. P<0.05 was considered to test for statistical significance difference.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of oral lesions meet the epithelial diagnostic criteria for mild to moderate grade OED
* No local area stimulate by residual root and crown, sharp cusp, poor restoration and biting cheek or lips
* Without the OCE treatment history by laser , radiation or chemical
* Be able to Sign the informed consent

Exclusion Criteria:

* Histopathological diagnosis of oral lesions do not meet the epithelium of mild to moderate dysplasia diagnostic criteria; histological diagnosis of severe grade OED or malignant disease
* Pregnancy or breast-feeding women
* Serious heart, lung, liver , kidney and other systemic diseases
* local area stimulate by residual root and crown, sharp cusp, poor restoration and biting cheek or lips
* OED treatment history by LASER, radiotherapy, or chemotherapy
* Tumor and psychiatric patients
* Patients are unable to cooperate

Ages: 25 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 180 patients with mild or moderate oral epithelial dysplasia were selected. 81 of them were from Peking University of Stomatology and 68 were from Capital Medical University School of Stomatology and other 31 were from Fourth Military Medical University School of Stomatology.All of the patients with OED had been diagnosed pathologically by at least two senior pathologists using the criteria from '2005 WHO Classification System' and The oral tissue pathology diagnostic criteria (oral histopathology Edition Sixth).All cases involved primary lesions without any LASER, radiation therapy or chemotherapy.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2009-02; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Cancer rate in patients with oral epithelial dysplasia containing or NOT containing p16 methylation | frome 3 months to 63 months
  152 participants were p16 methylated informative. 29 participants were NOT informative because enough DNA was not extracted from their paraffin slides.
  Among these informative cases, oral specimens from 48 patients were p16 methylation positive and 104 patients were p16 methylation negative. The cancer rate in the p16 methylation positive patients during the followup period will be compared with that in the p16 methylation negative patients statistically.

CONTACTS AND LOCATIONS:
Overall Officials: Dajun Deng, MD, Principal Investigator — Peking University

REFERENCES:
- See also: Peking University — http://www.pku.edu.cn